CLINICAL TRIAL: NCT03532022
Title: An Open-label, Randomized, Titration-blinded, Phase III Study of Efficacy, Safety and Tolerability Of Chronocort® Compared With Standard Glucocorticoid REeplacement Therapy in the Treatment of Participants Aged 16 Years and Over With Congenital Adrenal Hyperplasia
Brief Title: Open-label Comparison of Chronocort® Versus Standard Glucocorticoid Replacement Therapy
Acronym: RESTORE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Protocol re-design required following EU Phase III results
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-007
Record Dates: First submitted 2018-04-18; First posted 2018-05-22 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Standard of Care; Hydrocortisone; Dexamethasone; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chronocort (Experimental): Hydrocortisone modified release capsules - Chronocort®. 66 subjects will be randomised to this group using an interactive web response system (IWRS).
  Interventions: Drug: Chronocort®
- Standard Care (Active Comparator): Subjects participating in this arm will continue to receive their normal, standard care (hydrocortisone, dexamethasone, prednisone, prednisolone) once enrolled on the study. 66 subjects will be randomised to this arm using an interactive web response system (IWRS).
  Interventions: Drug: Standard Care

INTERVENTIONS:
Drug: Chronocort® — Hydrocortisone modified release capsules - 5mg, 10mg and 20mg.
  Other Names: Hydrocortisone modified release capsules
  Arms: Chronocort
Drug: Standard Care — The subject's standard care regimen upon entering the study; this could consist of hydrocortisone, dexamethasone, prednisone or prednisolone.
  Other Names: Hydrocortisone; Dexamethasone; Prednisone; Prednisolone
  Arms: Standard Care

SUMMARY:
This study is an open-label, randomised, titration-blinded, parallel arm, multicenter study to compare twice daily Chronocort® with standard care in participants with Congenital Adrenal Hyperplasia (CAH). This study will be conducted in the USA.

DETAILED DESCRIPTION:
It will compare the efficacy, safety and tolerability of twice daily Chronocort® with standard care (using the participant's usual individualized standard glucocorticoid regimen) over a treatment period of 52 weeks in participants aged 16 years and over with known CAH due to 21-hydroxylase deficiency (classic CAH) diagnosed in childhood with documented (at any time) elevated 17-OHP or A4 and currently treated with hydrocortisone, prednisone, prednisolone or dexamethasone (or a combination of the aforementioned glucocorticoids).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply (note: if a participant fails to meet an inclusion criterion, re-screening is permitted if the Investigator considers that the circumstances leading to screening failure will not be relevant when the participant is re-screened at a later time):

Age

1. Participant must be aged 16 years or older at the time of signing the informed consent.
2. In participants aged <18 years, height velocity must be less than 2 cm in the last year and puberty must be completed.

   Type of Participant and Disease Characteristics
3. Participants with known CAH due to 21-hydroxylase deficiency (classic CAH) diagnosed in childhood with documented (at any time) elevated 17-OHP or A4 and currently treated with hydrocortisone, prednisone, prednisolone or dexamethasone (or a combination of the aforementioned glucocorticoids).

   Sex
4. Male and female participants

   1. Male participants:

      - A male participant must agree to use contraception as detailed in Section 10.4 of this protocol during the treatment period and refrain from donating sperm during this period.
   2. Female participants:

      * A female participant is eligible to participate if she is not pregnant (Section 10.4), not breastfeeding, and at least one of the following conditions applies:

   i. Not a woman of childbearing potential (WOCBP) as defined in Section 10.4. OR ii. A WOCBP with a negative pregnancy test at entry into the study who agrees to follow the contraceptive guidance in Section 10.4 during the treatment period.

   Note: females presenting with oligomenorrhea or amenorrhea who are aged ≤55 years should be considered potentially fertile and therefore, as well as undergoing pregnancy testing like all other female participants, will be expected to be using an acceptable method of contraception which should have been ongoing for ≥90 days prior to the study.

   Informed Consent
5. Capable of giving signed informed consent as described in Section 10.1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply (note: if a participant meets an exclusion criterion, re-screening is permitted if the Investigator considers that the circumstances leading to screening failure will not be relevant when the participant is re-screened at a later time):

Medical Conditions

1. Clinical or biochemical evidence of hepatic or renal disease e.g. creatinine > 2 times the upper limit of normal (ULN) or elevated liver function tests (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >2 times the ULN).
2. History of bilateral adrenalectomy.
3. History of malignancy (other than basal cell carcinoma successfully treated >26 weeks prior to entry into the study).
4. Participants who have type 1 diabetes or any participant who is receiving insulin.
5. Participants with any other significant medical or psychiatric conditions that in the opinion of the Investigator would preclude participation in the study.

   Prior/Concomitant Therapy
6. Participants on regular daily oral steroids for any indication other than CAH. Note: a participant should not be given any steroids (even on an irregular basis) within 5 days of a study visit. If there is a medical need for steroid treatment within this time frame then the visit should be postponed until a 5-day interval has elapsed.
7. Co-morbid condition requiring daily administration of a medication or consumption of any material that interferes with the metabolism of glucocorticoids (examples provided at http://medicine.iupui.edu/clinpharm/ddis/clinical-table/).
8. Participants who are receiving <10 mg hydrocortisone dose at baseline or the hydrocortisone dose equivalent.

   Prior/Concurrent Clinical Study Experience
9. Participation in another clinical study of an investigational or licensed drug or device within the 12 weeks prior to screening or during the study.
10. Inclusion in any natural history or translational research study that would require evaluation of androgen levels during the study period outside of this study protocol assessments.
11. Participants who have previously been exposed to Chronocort in studies DIUR-003, DIUR-005 or DIUR-006.

    Other Exclusions
12. Participants who routinely work night shifts and so do not sleep during the usual night-time hours.
13. Participants unable to comply with the requirements of the protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2021-07-09 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of Chronocort® versus standard care in terms of responder rate. | 52 weeks
  The proportion of participants after 52 weeks of treatment in the Chronocort® and standard care treatment groups achieving biochemical control. Participants with 17 OHP and A4 in the optimal (for 17-OHP) and reference range (for A4) at both timepoints of 09:00 and 13:00 hours will be classified as 'in biochemical control'; if at least one of these measurements is outside of the optimal (for 17-OHP) or reference range (for A4) they will be classified as 'not in biochemical control'.

SECONDARY OUTCOMES:
Impact of both treatments on markers of fertility. | Weeks 26 & 52
  Proportion of participants who are "responders" at Weeks 26 and 52 i.e. restoration of menses/more regular menses in women (patient diary used to record menstrual cycle details in pre menopausal women who have not had a hysterectomy and are not using hormonal contraception), and luteinizing hormone (LH) in men that was outside the normal range at baseline but moves to within the normal range during the study
Impact of both treatments on hirsutism in female participants. | Weeks 26 & 52
  Change in hirsutism will be assessed at Weeks 26 and 52 using a 10 cm VAS ranging from 'No Symptoms' to 'Very Severe Symptoms' which will be completed by the participant.
Impact of both treatments on acne. | Weeks 26 & 52
  Change in acne assessed at Weeks 26 and 52 using a 10 cm visual analogue scale (VAS) ranging from 'No Symptoms' to 'Very Severe Symptoms' which will be completed by the participant.
Impact of both treatments on glycated hemoglobin (HbA1c) levels. | Weeks 26 & 52
  Change from baseline to Weeks 26 and 52 in glycated hemoglobin (HbA1c) levels.
Impact of both treatments on waist circumference (in centimetres). | Weeks 26 & 52
  Change from baseline to Weeks 26 and 52 in waist circumference (cm).
Impact of both treatments on body weight (in kilograms). | Weeks 26 & 52
  Change from baseline to Weeks 26 and 52 in body weight (kg).
Impact of both treatments on quality of life (QoL) using SF-36® total score and the sub-domain of vitality. | Weeks 26 & 52
  Change from baseline to Weeks 26 and 52 in Quality of Life using SF-36® total score and the score for the vitality sub-domain.
Impact of both treatments on Quality of Life using Multidimensional Assessment of Fatigue (MAF). | Weeks 26 & 52
  Change from baseline to Weeks 26 and 52 in Quality of Life using Multidimensional Assessment of Fatigue (MAF).
Impact of both treatments on Quality of Life using EQ-5D™. | Weeks 26 & 52
  Change from baseline to Weeks 26 and 52 in Quality of Life using EQ-5D™.
Safety and tolerability of Chronocort® relative to standard care | 52 weeks
  Incidence of clinical AEs, with a particular focus on adrenal crises.
The need for additional glucocorticoid doses | 52 weeks
  Use of immediate release hydrocortisone from the sick day packs or use of any additional glucocorticoid treatment during the study.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - Red blood cell count and platelet count | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare red blood cell and platelet counts (absolute values) between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - haemaglobin | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare haemaglobin concentrations (g/dL) between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - haematocrit | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare haematocrit levels (ratio of red blood cells to total blood volume) between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - mean corpuscular volume (MCV) | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare mean corpuscular volumes (volume of red blood cells) between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - mean cell haemoglobin (MCH) | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare mean cell haemoglobin concentrations between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - mean cell haemoglobin concentration (MCHC) | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare mean cell haemoglobin concentrations (as measured by dividing haematocrit by blood haemoglobin levels) between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - Red cell distribution width (RDW) | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare Red cell distribution width (measured in micrometres) between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of routine safety haematology assessments - White blood cell count with differential (absolute and %): Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Routine haematology assessments to compare average White blood cell counts (Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils) with differentials (absolute count and %) between the Chronocort arm and Standard Care arm.
Safety of Chronocort® compared to standard care by assessment of physical examinations. | Baseline (Day 1), Week 26 & Week 52
  Safety of Chronocort® compared to standard care as measured by the incidence of abnormal findings identified during physical examinations. The physical examination will include, at a minimum, assessments of the cardiovascular, respiratory, gastrointestinal and neurological systems for the purpose of safety monitoring and to determine subject eligibility. Investigators should pay special attention to clinical signs related to previous serious illnesses. Abnormal findings are recorded in the eCRF and are assessed for their clinical significance.
Safety of Chronocort® compared to standard care by assessment of vital signs - Blood pressure | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Systolic and diastolic blood pressure will be measured (in mmHg - millimetres of mercury) at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of vital signs - Heart rate | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Heart rate will be measured (in beats per minute) at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of vital signs - Respiratory rate | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Respiratory rate will be measured (in breaths per minute) at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of vital signs - Oral body temperature | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Oral body temperature (measured in Celsius) will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - Specific gravity | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Specific gravity of urine (concentration of solutes) will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - pH | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Urine pH (potential of hydrogen - molar concentration of hydrogen ions) will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - Glucose | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Urine glucose concentrations will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - Proteins | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Urine protein concentrations will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - Blood | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Concentration of blood molecules in urine will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - Ketones | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Urine ketone concentrations will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - Bilirubin | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Urine bilirubin concentrations will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of urinalysis - Urobilinogen by dipstick | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  Urobilinogen concentrations will be measured at each visit for safety monitoring purposes.
Safety of Chronocort® compared to standard care by assessment of electrocardiogram (ECG). | Baseline (Day 1), Week 2, Week 6, Week 12, Week 26, Week 39 & Week 52
  A single 12-lead ECG will be recorded using an ECG machine that automatically calculates and measures PR, QRS, QT and QTc intervals (in milliseconds and voltage). ECG measurements should be preceded by 10 minutes of rest (semi-supine) in a quiet area. ECGs will be read at sites by the local investigator and any abnormal findings recorded in the eCRF and the original ECG source notes stored in the participant's source notes.

CONTACTS AND LOCATIONS:
Locations (1):
- Diabetes and Endocrinology Consultants PC, Morehead City, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No